CLINICAL TRIAL: NCT01797731
Title: Conventional Tibial Extramedullary Alignment System Versus a Hand-Held, Surgical Navigation System for Tibial Component Placement in Total Knee Arthroplasty: A Randomized, Controlled Trial
Brief Title: Conventional Alignment System Versus Surgical Navigation System in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10137
Record Dates: First submitted 2013-02-07; First posted 2013-02-22 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Orthalign; KneeAlign; Total Knee Replacement; Total Knee Arthroplasty; Degenerative joint disease; Osteoarthritis; Unilateral
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional System (Active Comparator): Conventional tibial extramedullary alignment system used by surgeon during surgery.
  Interventions: Device: Conventional tibial extramedullary alignment system
- KneeAlign System (Experimental): Digital hand-held surgical navigation system for tibial component placement used by surgeon during surgery.
  Interventions: Device: Digital hand-held surgical navigation system

INTERVENTIONS:
Device: Digital hand-held surgical navigation system — Digital hand-held surgical navigation system used for tibial component placement in total knee arthroplasty
  Other Names: KneeAlign; OrthAlign
  Arms: KneeAlign System
Device: Conventional tibial extramedullary alignment system — This is the standard of care for total knee arthroplasty.
  Arms: Conventional System

SUMMARY:
This is a randomized, controlled, blinded prospective study comparing the use of the usual cutting guides with a palm-sized digital surgical navigation system in unilateral total knee arthroplasty. Analysis of pre- and post-operative X-rays will be used to compare alignment of the tibial (shinbone) implant components. The investigators expect that the FDA-approved hand-held surgical navigation device will increase the accuracy and precision of the tibial cut by telling the surgeon the exact position of the cutting block before the surgeon makes the cut, allowing minor adjustments to be made. The investigators expect the conventional device to take less time to use, but that this difference will decrease as the surgeon becomes more familiar with the device. The investigators expect the intraoperative measurements acquired by the KneeAlign system to strongly correlate with the radiographic alignments measured postoperatively.

DETAILED DESCRIPTION:
Medical records, private office charts, and electronic medical records will be utilized by the co-investigators to review data on patients who fit the previously stated inclusion criteria. Demographic data including age, gender, height (cm), and weight (kg) will be collected. Preoperative, standing anteroposterior hip-to-ankle radiographs will be measured for the lower extremity mechanical axis, the tibiofemoral anatomic alignment, and the distal femoral and proximal tibial anatomic angles. Intraoperative time measurements for use of both the conventional extramedullary alignment guide, and the KneeAlignTM system will be measured and recorded. The time required to utilize each alignment guide will be measured in seconds, starting from the time at which the surgeon is handed the alignment guide (KneeAlignTM or conventional, extramedullary), to the time at which the surgeon is handed the oscillating saw to make the tibial cut. Of note, no intraoperative alignment measurements are required or will be recorded for the conventional, extramedullary systems, while intraoperative alignments reported by the KneeAlignTM system will be recorded when the KneeAlignTM device is used. In addition, regarding the use of conventional, extramedullary tibial guides, each surgeon will utilize the guide (regardless of manufacturer) which they currently use most frequently when performing a total knee arthroplasty. While there may be minimal differences with regards each of the surgeon's conventional guides, they are all essentially the same with regards to utilizing an extramedullary rod for alignment of the tibial resection.

Currently, a total knee replacement requires an average tourniquet time of 30-50 minutes depending on the surgeon. We estimate an approximate increase in total tourniquet time of 5-6 minutes when using the hand-held surgical navigation system.

For each procedure (either KneeAlignTM or conventional, extramedullary guides), after making the initial cut, if at any point in the procedure the surgeon re-cuts the tibia, they will be asked a series of questions postoperatively as to why they re-cut the tibia as part of the data collection. These questions will include:

1. Did you re-cut the tibia because you thought more varus or valgus was required?
2. Did you re-cut the tibia to increase or decrease the posterior slope?
3. Did you re-cut the tibia to increase the amount of bone resected?
4. Were you happy with the overall tibial alignment? Postoperative radiographs will be obtained as part of each surgeon's postoperative protocol, and will include a standing anteroposterior hip-to-ankle radiograph and a standing lateral knee-to-ankle radiograph, from which the lower extremity mechanical axis, the tibiofemoral anatomic alignment, the tibial component mechanical alignment, and the tibial component posterior slope will be measured.

This study has the potential to provide significant information regarding the clinical accuracy and precision of the KneeAlignTM system compared to that of conventional, extramedullary alignment systems. If mechanical and tibial mechanical alignment is significantly improved with the use of the KneeAlignTM system, this may encourage surgeons to utilize this device to improve postoperative alignment in total knee arthroplasty. In addition, surgeon's may find this type of hand-held system more user-friendly (in contrast to a large console, computer-assisted surgical system), and this may stimulate future investigations into similar devices for femoral component alignment, and also total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* a history of osteoarthritis, rheumatoid arthritis, or post-traumatic arthritis
* patients who have been indicated for a primary, posterior-stabilized, total knee arthroplasty
* patients have had a preoperative standing anteroposterior hip-to-ankle radiograph and standing lateral knee-to-ankle radiographs

Exclusion Criteria:

* patients with proximal tibial defects requiring either a metal or allograft augment
* inadequate radiographic studies as required by the study protocol
* if they do not receive a total knee arthroplasty, or receive a unicondylar arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mayman, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Result] Nam D, Weeks KD, Reinhardt KR, Nawabi DH, Cross MB, Mayman DJ. Accelerometer-based, portable navigation vs imageless, large-console computer-assisted navigation in total knee arthroplasty: a comparison of radiographic results. J Arthroplasty. 2013 Feb;28(2):255-61. doi: 10.1016/j.arth.2012.04.023. Epub 2012 Jun 14. PMID 22704226
- [Result] Nam D, Jerabek SA, Cross MB, Mayman DJ. Cadaveric analysis of an accelerometer-based portable navigation device for distal femoral cutting block alignment in total knee arthroplasty. Comput Aided Surg. 2012;17(4):205-10. doi: 10.3109/10929088.2012.689335. Epub 2012 Jun 8. PMID 22681247
- [Result] Nam D, Nawabi DH, Cross MB, Heyse TJ, Mayman DJ. Accelerometer-based computer navigation for performing the distal femoral resection in total knee arthroplasty. J Arthroplasty. 2012 Oct;27(9):1717-22. doi: 10.1016/j.arth.2012.02.007. Epub 2012 Mar 21. PMID 22440228
- [Result] Nam D, Dy CJ, Cross MB, Kang MN, Mayman DJ. Cadaveric results of an accelerometer based, extramedullary navigation system for the tibial resection in total knee arthroplasty. Knee. 2012 Oct;19(5):617-21. doi: 10.1016/j.knee.2011.09.008. Epub 2011 Oct 26. PMID 22032868
- [Result] Nam D, Jerabek SA, Haughom B, Cross MB, Reinhardt KR, Mayman DJ. Radiographic analysis of a hand-held surgical navigation system for tibial resection in total knee arthroplasty. J Arthroplasty. 2011 Dec;26(8):1527-33. doi: 10.1016/j.arth.2011.01.012. Epub 2011 Mar 11. PMID 21397455

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional System | KneeAlign System
Started | 50 | 50
Completed | 47 (3 were excluded due to not having proper radiographs for adequate follow up) | 47 (3 excluded due to not having proper radiographs for adequate follow up)
Not Completed | 3 | 3
Not completed — Didn't have proper radiographs required | 3 | 3

BASELINE CHARACTERISTICS:
Population: A sample size of 47 patients in each cohort would provide appropriate power (beta level = 0.80, alpha level = 0.05) to detect a 20% improvement in accuracy between the two groups (i.e. a 20% decrease or increase in the number of "outliers").
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional System | KneeAlign System | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 17 | 44
  >=65 years | 20 | 30 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (10.1) | 67.1 (7.5) | 66.12 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 29 | 49
  Male | 27 | 18 | 45

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Tibial Component Alignment
Description: The primary outcome will be the number of patients (percentage of patients) that met a predetermined criteria for Alignment as defined by within 2° of perpendicular to the tibial mechanical axis or 2° of a 3° posterior slope, postoperative tibial component alignment (mechanical varus/valgus, and posterior slope) as measured on postoperative standing anteroposterior hip-to-ankle radiographs, and standing, lateral knee-to-ankle radiographs, respectively.
Time Frame: 6 weeks after surgery
Measure: Number; unit: percentage of participants
Arm/Group | Conventional System | KneeAlign System
Number analyzed (Participants) | 47 | 47
percentage of participants | 68.1 | 95.7

2. Secondary Outcome: Time Required to Utilize System
Description: The amount of time required to utilize conventional, tibial extramedullary alignment guides versus the KneeAlignTM system, which will be recorded intraoperatively.
Time Frame: Minutes during surgery ( Estimated time per surgery 1 hour)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Conventional System | KneeAlign System
Number analyzed (Participants) | 50 | 50
seconds | 289.92 (125.34) | 70.58 (28.14)

ADVERSE EVENTS:
Arm/Group | Conventional System | KneeAlign System
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes